CLINICAL TRIAL: NCT05269459
Title: Safety and Efficacy of Cannabidiol (CBD) for Symptoms of Post-Traumatic Stress Disorder (PTSD) in Adults Using Liquid StructureTM Formulation (NantheiaTM ATL5).
Brief Title: Safety and Efficacy of Cannabidiol (CBD) for Symptoms of PTSD in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Ananda Scientific Inc (Unknown); University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0159-22-FB
Record Dates: First submitted 2022-02-24; First posted 2022-03-08 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: PTSD
Keywords: PTSD; CBD; Nantheia ATL5; Quality of Life; Mobility; Tolerability; Cannabidiol
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Double-Blind Placebo Controlled Study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and study personnel are blinded to treatment assignment. Randomization will occur in blocks based on self-reported marijuana use (yes/no). Randomization schedule will be provided by the statistician to the research pharmacist for study drug dispensing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cannabidiol Administered as Nantheia ATL5 Group (Experimental): Cannabidiol (CBD) as Liquid Structure Formulation Nantheia ATL5 400mg will be administered twice a day in 100mg softgel capsules to CBD Group. Each 100mg softgel contains 10% CBD.
  Interventions: Drug: Cannabidiol Administered as Nantheia ATL5
- Placebo Group (Placebo Comparator): Matching placebo capsules will be administered twice a day to Placebo Group.
  Interventions: Drug: Placebo
- Control Group (No Intervention): Baseline data collection only will be collected from Control group.

INTERVENTIONS:
Drug: Cannabidiol Administered as Nantheia ATL5 — Participants will take 4 gel capsules twice daily containing 100mg of Nantheia ATL5.
  Other Names: CBD
  Arms: Cannabidiol Administered as Nantheia ATL5 Group
Drug: Placebo — Participants will take 4 matching gel capsules twice daily containing no active drug.
  Other Names: PBO
  Arms: Placebo Group

SUMMARY:
Post-traumatic stress disorder (PTSD) is a psychiatric disorder than may develop following a traumatic event including serious incidents, natural or human-caused disasters, violence, death of a loved one, receipt of traumatic news, or serious illness/hospitalization. While half of US adults experience trauma in their lifetime, most do not develop PTSD. However, those who do develop the disorder may have significant impairments and risk for functional dysfunction across multiple domains. While short term symptoms are the most common, some individuals develop chronic PTSD. These individuals may experience frightening and intrusive thoughts and memories of the event (flashbacks), have sleep disturbances, feel numb or detached, and be easily startled (hypervigilance).

This trial is a double-blind placebo controlled study of cannabidiol (CBD) for symptoms of PTSD in adults using liquid structure Formulation (Nantheia ATL5). Participants complete three weeks of baseline data collection including assessments of activity and sleep. Intervention is Nantheia ATL5 or placebo. Dose is initiated at 400mg BID and maintained over 8 weeks. Standardized symptom profile measurements, clinician assessments, laboratory testing, collection of inflammatory biomarkers, and suicide screening is completed throughout. Age- and gender-matched healthy population participants are enrolled and complete baseline data collection only. All participants may complete optional functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a psychiatric disorder than may develop following a traumatic event including serious incidents, natural or human-caused disasters, violence, death of a loved one, receipt of traumatic news, or serious illness/hospitalization. While half of US adults experience trauma in their lifetime, most do not develop PTSD. However, those who do develop the disorder may have significant impairments and risk for functional dysfunction across multiple domains. While short term symptoms are the most common, some individuals develop chronic PTSD. These individuals may experience frightening and intrusive thoughts and memories of the event (flashbacks), have sleep disturbances, feel numb or detached, and be easily startled (hypervigilance).

This trial is a single-site phase II, double-blind, placebo-controlled study of Nantheia ATL5 to study symptoms of Post-Traumatic Stress Disorder (PTSD) in adults. Participants will meet criteria for PTSD using the Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Clinical Assessment of Pragmatics (CAPs-5) of ≥ 27. Suicidality is assessed using the Columbia Suicide Severity Rating Scale-Revised (CSSRS-R) at all study visits. Baseline psychopharmacotherapy and/or psychotherapy must be stable (unchanged) for 4 weeks prior to enrollment and should remain unchanged during study treatment. Effects of Nantheia ATL5 on self-reported quality of life (overall and health-related); functional status measurements of personal mobility and risk, and sleep dysfunction; neurobiological biomarkers of threat response (optional functional magnetic resonance imaging: fMRI), and serum inflammatory biomarkers (hs-CRP) implicated in PTSD pathophysiology will be assessed. Efficacy and tolerability will be assessed throughout intervention. Serum pregnancy (for participants of child bearing potential), urine drug screening, complete blood count (CBC), and Comprehensive Metabolic Panel are completed at every on-site visit. Optional consent will be sought from all PTSD and healthy population participants who agree to complete the functional magnetic resonance imaging (fMRI) procedures and providing an additional sample of blood to store for future unspecified research. Baseline characteristics of participants with PTSD will be evaluated overall and relative to participants without PTSD (healthy population) during a 3-week baseline period prior to randomization [Nantheia ATL5 or placebo (PBO)]. Healthy population participants will complete the study at end of baseline and participants with PTSD will be randomized 1:1 to Nantheia ATL5 or placebo (PBO). Study drug dose is initiated at 400mg BID and maintained for 8 weeks. Study drug is then withdrawn, and one week later safety measures including laboratory testing, assessment of AE's and CSSRS-R are repeated.

ELIGIBILITY:
Inclusion Criteria All Participants

* Ability and willingness to provide informed consent
* Stated willingness to comply with all study procedures and availability for duration of the study
* Aged 21-65 years
* Able to read and communicate in English
* Tetrahydrocannabinol (THC) use less than 3 days per week

PTSD Participants

* Meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for a current diagnosis of Post-Traumatic Stress Disorder (PTSD) on the Mini-Mental State examination (MMS), with symptoms present for at least 1 month
* Clinician administered Clinical Assessment of Pragmatics (CAPs) score ≥27 at study enrollment and start of Cannabidiol (CBD) observation
* Stable psychopharmacologic and/or psychotherapeutic intervention for 4 weeks prior to enrollment

Exclusion Criteria All Participants

* Current use of prescribed or commercially available CBD products, including Epidiolex®
* Suicidal ideation (as defined by answer of "yes" to item 4 or 5 on the baseline Columbia Suicide Severity Rating Scale (C-SSRS) or attempt within 6 months prior to enrollment)
* Cognitive impairment in the clinical judgment of the investigator that would impact ability to complete study assessments or confound study results (e.g., neurodegenerative condition or other)
* Meets criteria for substance or alcohol use disorder of moderate or greater severity within 6 months prior to study enrollment based on the Mini-Mental State examination (MMS); nicotine dependence permitted
* Self-reported cannabis use on > 3 days/week starting 4 weeks prior to enrollment
* Positive urine drug screen for illicit substances other than cannabis
* Pregnant [confirmed by serum human chorionic gonadotropin (hCG) test], or breastfeeding
* Co-morbid medical conditions or concomitant treatments that may adversely impact ability to participate in the trial in the clinical judgment of the investigator [e.g., significant immunosuppression due to active chemotherapy, recent organ transplant, uncontrolled diabetes, glomerular filtration rate (GFR) < 25ml/min or on dialysis, recent acute myocardial infarction (MI), Class IV heart failure, or taking any high-risk drugs for drug-drug interactions]
* Treatment with another investigational drug or other intervention within 3 months prior to enrollment
* History of psychosis (schizophrenia, schizophreniform disorder, schizoaffective disorder, or substance induced psychosis), active bipolar disorder, or borderline personality disorder diagnosed by a mental health professional
* History of open head injury
* Self-report of exposure to trauma within 30 days prior to enrollment
* Active military service in the 30 days prior to enrollment
* Inpatient psychiatric hospitalization within 6 months prior to enrollment
* Seizure in the last 6 months
* Use of concomitant anti-viral human immunodeficiency virus (HIV) medications (PrEP permitted)

Control Participants

* History of diagnosed PTSD
* Pregnant (self-reported) or breastfeeding

Participants who consent to functional magnetic resonance imaging (fMRI) procedures

* Claustrophobia, pregnancy, or any condition (e.g., significant hearing difficulties) that would preclude MRI scanning, in the clinical judgment of the investigator
* Presence of metal objects in or on the body (e.g., pacemakers, aneurysm clips, metallic prostheses, bone plates, braces, orthodontic devices, cochlear implants/hearing aids, non-removable piercings/implants or metallic-ink tattoos, or shrapnel fragments)
* Other confounding medical conditions (e.g., Tourette's or Tic Disorder) that would preclude MRI scanning, in the clinical judgement of the investigator

PTSD Participants

* Index trauma before age 18 and no other traumatic experiences which could relate/identify as part of PTSD
* History of allergic reaction or significant adverse events (AE) related to cannabis, CBD, or THC
* Currently involved in events giving rise to PTSD
* Alanine transaminase (ALT)/Aspartate transaminase (AST)/Bilirubin > 2 x upper limit of normal (ULN) at screening (abnormalities on the comprehensive metabolic panel or complete blood count deemed to be of clinical significance in the judgement of the investigator and clinical team will be evaluated in the clinical context of the participant's history and physical examination to determine eligibility and testing may be repeated if clinically appropriate at the discretion of the investigator)
* Refusal to use at least one form of birth control throughout study participation [including, but are not limited to, male or female condoms, diaphragm, or cervical cap (all with or without spermicide) abstinence, or hormonal/implanted birth control, e.g., pill, injection, intra-uterine device (IUD), implant] by participants who can become pregnant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic Stress Disorder Symptom Rating | Baseline and 8 weeks
  Structured clinician-administered rating of post-traumatic stress disorder (PTSD) symptoms' severity using the Diagnostic and Statistical Manual of Mental Disorders (DSM-5; CAPS-5) Scale. This instrument assesses 20 PTSD symptoms. Each symptom is scored 0 - 4, then symptom scores are totaled. Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Post-traumatic Stress Disorder Symptom Symptom Cluster Rating | Baseline and 8 weeks
  The cluster scores (symptom domains) are subscales of the CAPS-5 (outcome 1). The CAPS-5 has 20 items, each scored 0-4. The sum of items 1-5 represent cluster B (intrusion symptoms); items 6-7 represent cluster C (avoidance symptoms); items 8-14 represent cluster D (cognitions and mood symptoms); and items 15-20 represent cluster E (arousal and reactivity symptoms). Score ranges are: Cluster B 0-20, Cluster C 0-8, Cluster D 0-28, and Cluster E 0-24.
  The total of the cluster scores (B+C+D+E) is the total CAPS-5 score.
  Higher scores indicate greater symptom severity.
Post-traumatic Stress Disorder Symptom Rating (Self-reported) | Baseline and 8 weeks
  Self-reported rating of post-traumatic stress disorder (PTSD) symptom severity using the PTSD Checklist for DSM-5 (PCL-5). This instrument the 20 items corresponding to the DSM-5 symptom criteria for PTSD. Each item is scored 0 - 4, then symptom scores are totaled. Higher scores indicate greater symptom severity.
Clinical Global Impression Post-traumatic Stress Disorder - Severity | Baseline and 8 weeks
  Clinical Global Impression Post-traumatic Stress Disorder (PTSD) Symptom Severity (CGI-S) is the assessment by clinicians of the severity of PTSD symptoms based on their experience with adults with PTSD. The CGI-S is scored on a scale of 0 to 7 (0 is "not assessed," 1 is "very much improved and 7 is "very much worse.") Higher scores indicate Higher scores indicate more severe illness.
Clinical Global Impression - Improvement | Baseline and 8 weeks
  Clinical Global Impression-Improvement (CGI-I) is the assessment by clinicians of the degree of post-traumatic stress disorder (PTSD) symptom improvement based on their experience with the population. It is rated without regard for relatedness to study treatment. The CGI-I is rated on a scale of 0 to 7 (0 is "not assessed," 1 is "very much improved and 7 is"very much worse.") Higher scores indicate worsening of symptoms.
Anxiety Severity Rating | Baseline and 8 weeks
  Clinician-rated assessment of anxiety symptoms using the Hamilton Anxiety Rating Scale (HAM-A). This instrument assesses 14 psychic (mental agitation and psychological distress) and somatic (related physical complaints) anxiety items. Each item is scored from 0 - 4, then symptom scores are totaled. Higher scores indicate greater anxiety severity.
Depression Symptoms Rating | Baseline and 8 weeks
  Clinician-rated assessment of depressive symptoms using the Hamilton Depression Rating Scale (HAM-D). This instrument assesses mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Each item is scored on a 3 or 5 point scale, depending on the item, then item scores are totaled. Higher scores indicate greater depressive symptoms.
Global Functioning Disability Questionnaire | Baseline and 8 weeks
  Participant-reported assessment of global functioning (an individual's overall ability to cope with daily life and maintain social, occupational, and psychological well-being) using the Sheehan Disability Scale (SDS). This instrument assesses functional impairment in work/school, social life, and family/home life. Each area is scored 0 - 10, then area scores are totaled. Higher scores indicate greater functioning disability.
Quality of Life Health Survey | Baseline and 8 weeks
  Participant-reported measure of quality of life using the Short Form 36-Item Health Survey (SF-36). This instrument assesses physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Each item is scored 0 - 100, then item scores are totaled. Higher scores indicate greater better health.

OTHER OUTCOMES:
Treatment-Emergent Adverse Events | 8 weeks
  The number and frequency of spontaneously reported adverse events (any untoward or harmful medical occurrence) from enrollment through study completion will be recorded.
Hepatic Function Measured by Serum Alanine Aminotransferase | Baseline and 8 weeks
  The clinical measure of hepatic function as measured by serum alanine aminotransferase (ALT) will be determined at baseline and 8 weeks and reported for values of >3x the upper limit of normal (ULN).
Hepatic Function Measured by Serum Aspartate Aminotransferase | Baseline and 8 weeks
  The clinical measure of hepatic function as measured by serum aspartate aminotransferase (AST) will be determined at baseline and 8 weeks and reported for values of >3x the upper limit of normal (ULN).
Hepatic Function Measured by Serum Bilirubin | Baseline and 8 weeks
  The clinical measure of hepatic function as measured by serum bilirubin will be determined at baseline and 8 weeks and reported for values of >3x the upper limit of normal (ULN).
Events of Suicidality | 8 weeks
  The events of suicidality are assessed by the Columbia Suicide Severity Rating Scale-Revised (CSSRS-R) which are either 'yes' or 'no' responses. The number of events is the total number of 'yes' responses to items 2, 3, 4 or 5.
Serious Adverse Events | up to 12 weeks
  Number of serious adverse events (SAE), e.g., death (any death occurring within 30 days of the participant receiving study drug, regardless of continuation on the protocol), a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect, will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rizzo, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Association, A. P. (2013). Diagnostic and Statistical Manual 5. Washington D.C.: American Psychiatric Association.
- [Background] Association, A. P. (2017). Medications for PTSD. Retrieved from https://www.apa.org/ptsd-guideline/treatments/medications
- [Background] Stanciu CN, Brunette MF, Teja N, Budney AJ. Evidence for Use of Cannabinoids in Mood Disorders, Anxiety Disorders, and PTSD: A Systematic Review. Psychiatr Serv. 2021 Apr 1;72(4):429-436. doi: 10.1176/appi.ps.202000189. Epub 2021 Feb 3. PMID 33530732
- [Background] Wall MB, Pope R, Freeman TP, Kowalczyk OS, Demetriou L, Mokrysz C, Hindocha C, Lawn W, Bloomfield MA, Freeman AM, Feilding A, Nutt D, Curran HV. Dissociable effects of cannabis with and without cannabidiol on the human brain's resting-state functional connectivity. J Psychopharmacol. 2019 Jul;33(7):822-830. doi: 10.1177/0269881119841568. Epub 2019 Apr 23. PMID 31013455
- [Background] Sholler DJ, Schoene L, Spindle TR. Therapeutic Efficacy of Cannabidiol (CBD): A Review of the Evidence from Clinical Trials and Human Laboratory Studies. Curr Addict Rep. 2020 Sep;7(3):405-412. doi: 10.1007/s40429-020-00326-8. Epub 2020 Jul 25. PMID 33585159
- [Background] Marx BP, Lee DJ, Norman SB, Bovin MJ, Sloan DM, Weathers FW, Keane TM, Schnurr PP. Reliable and clinically significant change in the clinician-administered PTSD Scale for DSM-5 and PTSD Checklist for DSM-5 among male veterans. Psychol Assess. 2022 Feb;34(2):197-203. doi: 10.1037/pas0001098. Epub 2021 Dec 23. PMID 34941354
- [Background] Hurd YL. Leading the Next CBD Wave-Safety and Efficacy. JAMA Psychiatry. 2020 Apr 1;77(4):341-342. doi: 10.1001/jamapsychiatry.2019.4157. No abstract available. PMID 31940016
- [Background] Elsaid S, Kloiber S, Le Foll B. Effects of cannabidiol (CBD) in neuropsychiatric disorders: A review of pre-clinical and clinical findings. Prog Mol Biol Transl Sci. 2019;167:25-75. doi: 10.1016/bs.pmbts.2019.06.005. Epub 2019 Aug 28. PMID 31601406
- [Background] Andrewes DG, Jenkins LM. The Role of the Amygdala and the Ventromedial Prefrontal Cortex in Emotional Regulation: Implications for Post-traumatic Stress Disorder. Neuropsychol Rev. 2019 Jun;29(2):220-243. doi: 10.1007/s11065-019-09398-4. Epub 2019 Mar 14. PMID 30877420
- [Background] Babson KA, Sottile J, Morabito D. Cannabis, Cannabinoids, and Sleep: a Review of the Literature. Curr Psychiatry Rep. 2017 Apr;19(4):23. doi: 10.1007/s11920-017-0775-9. PMID 28349316
- [Background] Elms L, Shannon S, Hughes S, Lewis N. Cannabidiol in the Treatment of Post-Traumatic Stress Disorder: A Case Series. J Altern Complement Med. 2019 Apr;25(4):392-397. doi: 10.1089/acm.2018.0437. Epub 2018 Dec 13. PMID 30543451
- [Background] Hori H, Kim Y. Inflammation and post-traumatic stress disorder. Psychiatry Clin Neurosci. 2019 Apr;73(4):143-153. doi: 10.1111/pcn.12820. Epub 2019 Feb 21. PMID 30653780
- [Background] Jackson BN, Weathers FW, Jeffirs SM, Preston TJ, Brydon CM. The revised Clinician-Administered PTSD scale for DSM-5 (CAPS-5-R): Initial psychometric evaluation in a trauma-exposed community sample. J Trauma Stress. 2025 Feb;38(1):40-52. doi: 10.1002/jts.23093. Epub 2024 Aug 23. PMID 39176447